CLINICAL TRIAL: NCT06085885
Title: Evaluation of Factors Predicting Tinnitus Outcomes Following Cochlear Implantation
Brief Title: Tinnitus and Cochlear Implants
Acronym: TICIT
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Derek Hoare, Chief Investigator, University of Nottingham
Other Study IDs: 23004; 292855 (Other: IRAS project ID)
Record Dates: First submitted 2023-08-11; First posted 2023-10-17 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Cochlear Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cochlear implant recipients: This study involves no clinical interventions beyond cochlear implantation that will be already available to participants as part of their routine care pathway. Participants will undergo routine pre- and post-operative assessments as part of usual care.
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant — Cochlear implant

SUMMARY:
Objectives of this study are to (1) Determine whether there are meaningful changes in tinnitus outcomes following cochlear implantation in adults with bilateral severe-to-profound hearing loss, (2) Determine the prevalence, nature, and severity of tinnitus before cochlear implantation, (3) Determine the incidence, nature, and changes in severity of tinnitus following cochlear implantation, and (4) Explore associations between tinnitus and changes in hearing, psychological health, cochlear implantation-related factors, and quality of life in cochlear implant recipients with and without tinnitus.

Participants will be adults eligible to receive a unilateral cochlear implant on the National Health Service (NHS) in the United Kingdom (UK). Participants will undergo routine pre- and post-operative assessments as part of usual care, and complete online questionnaires before and after implantation to measure tinnitus and other health related factors. Mixed statistical methods will be used to characterise the sample and evaluate changes in the severity of tinnitus and patient-specific factors after implantation.

DETAILED DESCRIPTION:
Primary objective:

Determine whether there are meaningful changes in tinnitus outcomes following cochlear implantation in adults with bilateral severe-to-profound hearing loss.

Secondary objectives:

1. Determine the prevalence, nature, and severity of tinnitus before cochlear implantation.
2. Determine the incidence, nature, and changes in severity of tinnitus following cochlear implantation.
3. Explore associations between tinnitus and changes in hearing, psychological health, cochlear implantation-related factors, and quality of life in cochlear implant recipients with and without tinnitus.

Patient identification:

Providers of cochlear implantation services on the National Health Service in the United Kingdom.

The schedule of questionnaires will follow the schedule of routine clinical appointments as part of the cochlear implantation care pathway including a pre-operative baseline assessment, and five follow up assessments after the surgery to receive the cochlear implant, after the first cochlear implant activation appointment, and at routine 1-, 3- and 6-month appointments post-activation. The baseline questionnaires will require about 40 min to complete and follow up questionnaires about 15-30 min.

Detailed analyses will be specified prospectively in a study analysis plan developed by the study team. Data analyses will be conducted by the study team with support from medical statisticians at the National Institute for Health Research (NIHR) Nottingham Biomedical Research Centre (BRC). The software utilised for analyses may include Excel, SPSS, R or MATLAB. Mixed statistical methods will be used to characterise the sample and evaluate changes in the severity of tinnitus and patient-specific factors before and after implantation. Data analyses will include descriptive statistics, General/Generalised Linear Models (e.g., ANOVA, regression models) or non-parametric statistical methods where appropriate (e.g., Mann Whitney U test).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Determined to be eligible for unilateral cochlear implantation.
* Did not previously receive a cochlear implant in either ear.
* Sufficient written or spoken English to participate in study activities.
* Have access to internet or suitable device to complete online study questionnaires.
* Able to give informed consent.

Exclusion Criteria:

* Significant difficulties preventing independent completion of study activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe to profound hearing loss undergoing cochlear implantation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Tinnitus characteristics and associated medical and sociodemographic factors | Before cochlear implantation, two weeks after cochlear implantation, immediately after the activation of the cochlear implant, and one, three and six months after the activation of the cochlear implant
  The European School for Interdisciplinary Tinnitus Research Screening Questionnaire (ESiT-SQ). This is a case history questionnaire without a numerical scoring system.
Tinnitus impact | Before cochlear implantation, two weeks after cochlear implantation, immediately after the activation of the cochlear implant, and one, three and six months after the activation of the cochlear implant
  Tinnitus Functional Index (TFI). Maximum score: 250, higher score indicates greater tinnitus symptom severity
Patient health | Before cochlear implantation, two weeks after cochlear implantation, and one, three and six months after the activation of the cochlear implant
  Patient Health Questionnaire (PHQ-9) scores can range from 0 to 27 with a higher score indicating more severe symptoms
Anxiety | Before cochlear implantation, two weeks after cochlear implantation, and one, three and six months after the activation of the cochlear implant
  Generalised Anxiety Disorder Assessment (GAD-7) scored from 0 to 21, with a higher score indicating more severe anxiety
Insomnia | Before cochlear implantation, two weeks after cochlear implantation, and one, three and six months after the activation of the cochlear implant
  Insomnia Severity Index (ISI) scored 0 to 28 with a higher score indicating more severe insomnia
Life quality | Before cochlear implantation, two weeks after cochlear implantation, and one, three and six months after the activation of the cochlear implant
  EuroQol Quality of Life Questionnaire (EQ-5D-5L) scored from 0 to 100, with a lower score indicating worse health
Hearing function | Before cochlear implantation, two weeks after cochlear implantation, immediately after the activation of the cochlear implant, and one, three and six months after the activation of the cochlear implant
  Speech, Spatial and Qualities of Hearing (SSQ-12) questionnaire scored 0-120, with a higher score indicating better hearing ability

CONTACTS AND LOCATIONS:
Overall Officials: Derek J Hoare, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham Auditory Implant Programme, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No